CLINICAL TRIAL: NCT01724840
Title: Resection Suspension Arthroplasty With Interposition of GraftJacket Versus Tendon Interposition for Trapeziometacarpal Osteoarthritis: A Randomised Controlled Trial
Brief Title: GraftJacket Versus Tendon Interposition for Trapeziometacarpal Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Principal Investigator, Daniel Herren, MD, MHA, Schulthess Klinik
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GraftJacket01
Record Dates: First submitted 2012-11-01; First posted 2012-11-12 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthrosis of the Carpometacarpal Joint of the Thumb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GraftJacket (Experimental): GraftJAcket is used as interpositional material
  Interventions: Procedure: GraftJacket
- Tendon Interposition (Active Comparator): Flexor carpi radialis tendon is used as interpositional material
  Interventions: Procedure: Tendon Interposition

INTERVENTIONS:
Procedure: GraftJacket — Interposition with GraftJacket
  Arms: GraftJacket
Procedure: Tendon Interposition — Tendon Interposition with the FCR tendon
  Arms: Tendon Interposition

SUMMARY:
Studies at the shoulder, Achilles tendon and thumb show satisfactory results regarding the use of GaftJacket. Initial trials at the thumb show, that the GraftJacket can be safely and successfully used in TMC OA surgery and therefore represents an acceptable alternative for avoiding possible donor-site morbidity. However, there are no randomised controlled trials (RCT) in which the outcomes of using a tendon interposition or the GraftJacket are compared. Only with an RCT design it is possible to gain evidence about the advantages of one treatment method over another. The main objective of the study is the comparison between two surgical techniques for TMC OA: The resection interposition suspension arthroplasty using a part of the flexor carpi radialis tendon as interpositional material and using the GraftJacket as interpositional material.

DETAILED DESCRIPTION:
Besides the use of the flexor carpi radialis tendon, several materials can serve as the interposition tissue including Gore-Tex, silicone and other types of metal or polymer implants. The use of Gore-Tex, silicone and metal implants, have been shown to carry high complication rates secondary to synovitis and mechanical failure combined with poor patient outcomes. A study about a porcine collagen xenograft was terminated prematurely because of poor outcomes and adverse immunologic reactions.

Another option is using allograft, which is dermal or tendon tissue from another human donor such as the GraftJacket (Wright Medical Technology, Inc., Arlington, TN). This product is manufactured from donated cadaveric tissue that is treated to remove all cellular components while preserving the native collagen scaffold. It thus provides the strength and integrity of native autograft without the adverse immunologic response of traditional allograft. It is in compliance with the American Association of Tissue Banks guidelines for allograft material, and it is classified as human tissue for transplantation.

The GraftJacket shows high biocompatibility and the advantages compared to autograft are avoiding donor site morbidity as well as decreased surgical time.

GraftJacket has mainly being used for the repair of rotator cuff tears and Achilles tendons ruptures. No complications have been reported and patients showed significant improved outcomes compared with their preoperative conditions. Although all of the studies show methodological limitations due to the lack of a control group, these results show a great potential and warrant further investigations.

In contrast to the studies already conducted in the Achilles tendon and shoulder joint, there are only sparse data concerning other joints of the upper extremity such as the elbow and the hand. Treating TMC OA of Eaton stage ll, lll and lV with GraftJacket has only been reported in two studies. The patients under investigation reported significant pain relief, significant improvements regarding grip and key pinch strength, good ability to perform activities of daily living (ADL) and high satisfaction rates. No or only minimal postoperative complications such as paraesthesia which are not directly related to the GraftJacket have been reported. However, some limitations of these two studies have to be acknowledges. Both are observational studies without control group making it impossible to conclude if this approach is favourable compared to standard techniques.

ELIGIBILITY:
Inclusion criteria:

* All adult patients diagnosed for TMC OA
* willing to participate and provide informed consent

Exclusion criteria:

* Patients with rheumatoid arthritis,
* pregnant women,
* legal incompetent patients,
* persons with insufficient knowledge of the German language to complete the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Pain subscale of the Michigan Hand Questionnaire, 1 year following surgery | preOP, 6 weeks, 3, 6, and 12months post OP

SECONDARY OUTCOMES:
Secondary objectives are the comparison of the complications associated with the different surgical procedures as well as a cost-utility analysis. | preOP, 6 weeks, 3, 6, and 12months post OP

OTHER OUTCOMES:
Costs, Treatment satisfaction, objective and subjective function | preOP, 6 weeks, 3, 6, and 12months post OP

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Herren, MD, MHA, Principal Investigator — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Switzerland